CLINICAL TRIAL: NCT03772600
Title: Comparing Continuous With Flash Glucose Monitoring in Adults With Type 1 Diabetes
Acronym: ALERTT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, prof dr Pieter Gillard, Prof Dr, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S61830
Record Dates: First submitted 2018-12-05; First posted 2018-12-11 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Dexcom G6; FreeStyle Libre; time in range; continuous glucose monitoring; flash glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, double arm, open label, partial cross-over, parallel group clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexcom G6 (Experimental): Use a Dexcom G6 CGM for 36 months
  Interventions: Device: Dexcom G6 CGM
- FreeStyle Libre (No Intervention): Keep using their FreeStyle Libre for 6 months. Before the 6 month time point is reached, patients will wear a blinded Dexcom G6 for 28 days, together with their FreeStyle Libre.
  Cross-over to Dexcom G6 for 30 months.

INTERVENTIONS:
Device: Dexcom G6 CGM — Use of Dexcom G6
  Arms: Dexcom G6

SUMMARY:
The present study wants to compare the Dexcom G6® continuous glucose monitoring (CGM) system (experimental group) with the FreeStyle Libre flash glucose monitoring (FGM) system (control group).

The ALERTT1 trial will have three phases: a baseline, study, and extension phase.

During the baseline phase, eligible patients will be screened for in- and exclusion criteria, wear a blinded Dexcom G6® for 28 days, together with their FreeStyle Libre FGM system, and receive a uniform education moment.

In the study phase, patients will be randomized into two groups (1:1): the experimental group will use an unblinded Dexcom G6® CGM for 6 months, the control group will keep using the FreeStyle Libre FGM system for 6 months. Before the 6 month time point is reached, patients in the control group will wear a blinded Dexcom G6® CGM for 28 days, together with their FreeStyle Libre FGM.

In the extension phase, patients in the initial control group will start using unblinded Dexcom G6® for 30 months. The initial experimental group will keep using the unblinded Dexcom G6® for the next 30 months.

ELIGIBILITY:
Inclusion Criteria:

* signed ICF
* diagnosis of type 1 diabetes ≥6 months
* using FreeStyle Libre FGM system ≥6 months
* intensified insulin therapy/insulin pump therapy
* HbA1c ≤10%
* willing to wear the glucose monitoring device >80% of the time
* willing to download glucose monitoring data at regular intervals

Exclusion Criteria:

* non-type 1 diabetes participants or diagnosis <6 months
* participant with T1D not on insulin, or on non-intensified insulin therapy
* pregnancy or planning pregnancy within next 6 months
* severe cognitive dysfunction or other disease which makes sensor use difficult
* current treatment with drugs known to have significant interference with glucose metabolism, such as systemic corticosteroids, as judged by the investigator
* abnormal skin at the anticipated glucose sensor insertion sites (excessive hair, burn, inflammation, infection, rash, and/or tattoo)
* presence of concomitant pathology that might cause edema at the insertion sites (such as heart failure, liver failure, kidney failure defined as eGFR <30 mL/min [stage ≥4])
* beta-cell transplantation and c-peptide positive and/or under immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Difference in time in range (70-180 mg/dL) between the control and experimental group | 6 months
  measured by Dexcom G6

SECONDARY OUTCOMES:
Between group difference in time in clinically important hypoglycemia (<54mg/dL) | 6 months
  measured by Dexcom G6
Between group difference of HbA1c | 6 months
Between group difference in fear of hypoglycemia measured by the hypoglycemia fear survey | 6 months
Between group difference in time in hypoglycemia (<70 mg/dL) | 6 months
  measured by Dexcom G6
Between group difference in time in target (70-140 mg/dL) | 6 months
  measured by Dexcom G6
Between group difference in time in hyperglycemia (>180 mg/dL) | 6 months
  measured by Dexcom G6
Between group difference in time in clinically important hyperglycemia (>250 mg/dL) | 6 months
  measured by Dexcom G6
Composite endpoint: between group difference in number of patients with HbA1c <7% without episodes of severe hypoglycemia | 6 months
Between group difference in glycemic variability as measured by coefficient of variation [CV] | 6 months
  measured by Dexcom G6
Between group difference in glycemic variability as measured by standard deviation [SD] | 6 months
  measured by Dexcom G6
Between group difference in glycemic variability as measured by mean amplitude of glycemic excursions [MAGE] | 6 months
  measured by Dexcom G6
Between group difference in mean glucose concentration | 6 months
  measured by Dexcom G6
Between group difference in number of low glucose events (LGE) | 6 months
  LGE, measured by Dexcom G6, is defined as sensor glucose values ≤54 mg/dL for at least 15 minutes, preceded by at least 30 minutes with sensor glucose values >54 mg/dL
Between group difference in number of severe hypoglycemic episodes | 6 months
  reported by the participant
Between group difference in emotional distress due to diabetes measured by the problem areas in diabetes (PAID) questionnaire | 6 months
Between group difference in hypoglycemia awareness measured by the Clarke hypoglycemia awareness survey | 6 months
Between group difference in treatment satisfaction measured by the diabetes treatment satisfaction questionnaire (DTSQ) | 6 months
Between group difference in general quality of life measured by the SF-36 questionnaire | 6 months
Between group difference in number of patients having allergic reactions to the sensors | 6 months
  confirmed by a dermatologist

OTHER OUTCOMES:
Number of diabetes contacts which are not preplanned | 6 months
Resource utilization (cost material, use of extra adhesives) | 6 months
Number of severe adverse events | 6 months
Hospitalizations for severe acute diabetes complications (hypoglycemia and ketoacidosis) | 6 months
Work absenteeism due to diabetes | 6 months
Number of patients who stop using the Dexcom G6 CGM and the reason to stop | 6 months
Changes in time in range (70-180 mg/dL) | 36 months (extension phase)
  within-group change
Changes in time in target (70-140 mg/dL) | 36 months (extension phase)
  within-group change
Changes in time in hypoglycemia (<70 mg/dL) | 36 months (extension phase)
  within-group change
Changes in time in clinically important hypoglycemia (<54 mg/dL) | 36 months (extension phase)
  within-group change
Changes in time in hyperglycemia (>180 mg/dL) | 36 months (extension phase)
  within-group change
Changes in time in clinically important hyperglycemia (>250 mg/dL) | 36 months (extension phase)
  within-group change
Changes in time in glycemic variability, defined by coefficient of variation (CV) | 36 months (extension phase)
  within-group change
Changes in time in glycemic variability, defined by standard deviation (SD) | 36 months (extension phase)
  within-group change
Changes in time in glycemic variability, defined by mean amplitude of glycemic excursions (MAGE) | 36 months (extension phase)
  within-group change
Changes in time in number of low glucose events (LGE) (LGE is defined as sensor glucose values ≤54 mg/dL for at least 20 minutes, preceded by at least 30 minutes with sensor glucose values >54 mg/dL) | 36 months (extension phase)
  within-group change
Changes in HbA1c | 36 months (extension phase)
  within-group change
Changes in in emotional distress due to diabetes measured by the PAID questionnaire | 36 months (extension phase)
  within-group change
Changes in in hypoglycemia awareness measured by the Clarke hypoglycemia awareness survey | 36 months (extension phase)
  within-group change
Changes in treatment satisfaction measured by the DTSQ | 36 months (extension phase)
  within-group change
Changes in general quality of life measured by the SF-36 questionnaire | 36 months (extension phase)
  within-group change
Changes in in fear of hypoglycemia measured by the hypoglycemia fear survey | 36 months (extension phase)
  within-group change
Changes in hospitalizations for severe acute diabetes complications (hypoglycemia and ketoacidosis, expressed as admissions per patient year) | 36 months (extension phase)
  within-group change
Changes in work absenteeism (expressed as days of work absenteeism per patient year) | 36 months (extension phase)
  within-group change
Changes in number of severe hypoglycemic episodes (expressed as number of episodes per patient year) | 36 months (extension phase)
  within-group change
Number of patients who stop using the Dexcom G6® CGM and the reason to stop | 36 months (extension phase)
  within-group change

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (6):
  - Onze-Lieve-Vrouw Ziekenhuis Aalst, Aalst
  - Imeldaziekenhuis Bonheiden, Bonheiden
  - University Hospital Brussels, Jette
  - AZ Groeninge Kortrijk, Kortrijk
  - University Hospital Leuven, Leuven
  - University Hospital Antwerp, Wilrijk

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data can be shared with participating centers, based on research questions mentioned in this protocol or based on a new study protocol approved by the relevant ethical committees.

REFERENCES:
- [Derived] Visser MM, Van Muylder A, Charleer S, Isitt JJ, Roze S, De Block C, Maes T, Vanhaverbeke G, Nobels F, Keymeulen B, Mathieu C, Luyten J, Gillard P, Verhaeghe N. Cost-utility analysis of Dexcom G6 real-time continuous glucose monitoring versus FreeStyle Libre 1 intermittently scanned continuous glucose monitoring in adults with type 1 diabetes in Belgium. Diabetologia. 2024 Apr;67(4):650-662. doi: 10.1007/s00125-023-06084-2. Epub 2024 Jan 18. PMID 38236409
- [Derived] Visser MM, Charleer S, Fieuws S, De Block C, Hilbrands R, Van Huffel L, Maes T, Vanhaverbeke G, Dirinck E, Myngheer N, Vercammen C, Nobels F, Keymeulen B, Mathieu C, Gillard P. Effect of switching from intermittently scanned to real-time continuous glucose monitoring in adults with type 1 diabetes: 24-month results from the randomised ALERTT1 trial. Lancet Diabetes Endocrinol. 2023 Feb;11(2):96-108. doi: 10.1016/S2213-8587(22)00352-7. PMID 36702566
- [Derived] Visser MM, Charleer S, Fieuws S, De Block C, Hilbrands R, Van Huffel L, Maes T, Vanhaverbeke G, Dirinck E, Myngheer N, Vercammen C, Nobels F, Keymeulen B, Mathieu C, Gillard P. Comparing real-time and intermittently scanned continuous glucose monitoring in adults with type 1 diabetes (ALERTT1): a 6-month, prospective, multicentre, randomised controlled trial. Lancet. 2021 Jun 12;397(10291):2275-2283. doi: 10.1016/S0140-6736(21)00789-3. Epub 2021 Jun 2. PMID 34089660